CLINICAL TRIAL: NCT07066852
Title: Evaluation of the Effectiveness of Developmental Hip Dysplasia Screening in Risk Groups
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, KENAN ŞEN, Principal Investigator, Orthopedics and Traumatology Assistant, Ankara City Hospital Bilkent
Other Study IDs: DDHBilkent
Record Dates: First submitted 2024-11-12; First posted 2025-07-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Developmental Dysplasia of Hip
Keywords: acetabulardysplasia; screening; ultrasound; xray; developmentaldysplasiaofhip; PediatricOrthopedics
MeSH Terms: conditions — Hip Dislocation | interventions — X-Rays; Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- sample: we use one arm and one sample
  Interventions: Radiation: x ray; Diagnostic Test: ultrasound

INTERVENTIONS:
Radiation: x ray — we performed pelvis ap and frog leg x ray to child in 6 month and 1 age
Diagnostic Test: ultrasound — we will perform ultrasound in 6 week and 3 month

SUMMARY:
This study is a non-drug clinical trial.

Developmental dysplasia of the hip (DDH) encompasses a spectrum of hip developmental disorders, including dislocation, subluxation, and acetabular dysplasia. DDH is among the most prevalent hip conditions in infants. Dislocation is defined as the incomplete displacement of the hip joint, and residual dislocation due to DDH is associated with pain and severe osteoarthritis of the hip in young adulthood.

The progression of DDH is dynamic and may improve or worsen depending on various factors. The primary determinant of prognosis is the concentric reduction of the hip joint, with the femoral head needing to be reduced to allow for normal acetabular development.

DDH is the most common orthopedic condition in the neonatal period. According to the literature, the incidence is approximately 1:100 for dysplasia and 1:1000 for dislocation. However, estimates suggest that dislocation rates in Türkiye may reach 5-15:1000. DDH occurs six times more frequently in girls than boys and is more commonly observed in the left hip. Established risk factors for DDH include being a first-born girl, Caucasian race, positive family history, oligohydramnios, multiple pregnancies, in utero breech presentation, pes calcaneovalgus, metatarsus adductus, and torticollis.

Early detection and treatment of dislocation caused by DDH are associated with success rates exceeding 80%. However, diagnosis and treatment initiation after one year of age often result in variable outcomes. Literature indicates that clinical and sonographic evaluations may be normal at six weeks in breech patients-who are at significant risk for DDH-yet hip dysplasia may still develop in this population later. The investigators aim to contribute to existing literature by evaluating whether sonographic screening alone is sufficient or if additional screening methods are warranted for patients with identified DDH risk factors.

DETAILED DESCRIPTION:
Study Overview This study aims to evaluate the effectiveness of developmental dysplasia of the hip (DDH) screening in high-risk pediatric groups in Türkiye.

In Türkiye, all newborns undergo routine hip ultrasonography during the second month of life. If the results are normal, no further hip evaluations are typically performed. However, incidental detection of acetabular dysplasia in children-who later undergo pelvic anteroposterior (AP) X-rays for unrelated reasons-has raised concerns regarding the sufficiency of current screening protocols. Recent studies emphasize that hip development is a dynamic process, with the first 18 months being critical for early intervention. The timely detection of hip dysplasia is essential to minimize long-term physical and psychological burden on patients and healthcare systems. Undiagnosed cases often result in the need for total hip replacement surgery in adulthood. Accordingly, there is a need for a large-scale, prospective study to broaden and enhance the scope of DDH screening, both nationally and globally.

Study Population and Screening Protocol Participants will include all children born in the high-risk pregnancy ward at Ankara Bilkent City Hospital, selected via randomized sampling. After obtaining informed consent from families, hip ultrasonography will be performed six weeks postpartum using the Graf classification method. The screening will include Ortolani-Barlow maneuvers, Galeazzi sign assessment, swaddling practices, and evaluation of associated foot deformities. All sonographic assessments will be conducted by a single, qualified physician.

In cases where pathology is detected, treatment will be initiated in accordance with current medical guidelines. The Graf-based ultrasonography will be repeated at the third month, and follow-up clinical notes will be documented. At six months of age, pelvic AP and frog-leg lateral X-rays will be obtained. The acetabular index will be assessed using the Tönnis grading system, and any limitations in abduction will be recorded. At one year of age, follow-up X-rays will be performed to reassess the acetabular index and Tönnis grade, facilitating longitudinal monitoring of hip development during infancy.

Ethics and Statistical Evaluation Ethics approval for this study was granted by the Ethics Committee of Ankara Bilkent City Hospital (Board No. 1). Power analysis indicated a required sample size of 185 participants to achieve a statistical power of 0.95. This study will be conducted prospectively and analyzed using SPSS version 26.0. Findings will be reported to the Ministry of Health of Türkiye upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* All girls and boys of Turkish origin born in our hospital were included in our study.

Exclusion Criteria:

* Teratological hip diseases with neuromuscular disorders were excluded from our study. Parents who disrupted follow-up were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all children born in the high-risk pregnancy service at our hospital. Participants will be selected randomly, and their families will be informed about the study, providing consent for participation. The study aims to evaluate the effectiveness of developmental hip dysplasia (DDH) screening in high-risk groups in Turkey. Hip ultrasound will be performed six weeks after birth using the Graf method for screening purposes. This examination will include the Ortolani-Barlow test, Galeazzi sign, swaddling, and assessment of any accompanying foot deformities. All ultrasounds will be conducted by a single physician. If any pathology is detected, treatment will be initiated according to current literature. Follow-up evaluations will be conducted at three months, six months, and one year to monitor hip development and assess the acetabular index using Tönnis grading and abduction limitation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Acetabular Index Variation Measured by Tönnis Grading System | At 6 months and 1 year of age
  The change in acetabular index will be assessed using pelvic anteroposterior(AP) and frog-leg lateral x-rays. Measurements will be analyzed according to the classification system. The unit of measure will be degrees(°).

SECONDARY OUTCOMES:
Incidence of Pathological Findings on Graf Ultrasonography | At 6 weeks and 3 months after birth
  Rate of infants showing sonographic abnormalities(types 2b,2c,d,3,4) on graf uulrasound.Assessment will indclude morphological classification using Graf's criteria.Unit of measure:% of screened participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Safa Kapıcıoğlu, Proffesor, Study Director — Department of Orthopedics and Traumatology, Bilkent City Hospital, Ankara; Mehmet Safa Kapıcıoğlu, Proffesor, Principal Investigator — Department of Orthopedics and Traumatology, Bilkent City Hospital, Ankara
Locations (1):
- Department of Orthopedics and Traumatology, Bilkent City Hospital, Ankara, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I plan to share the code with famous journals as proof that I have done a prospective study. In addition, since this study means 1-year hip follow-up of 340 children and there is no follow-up of this size, I want it for proof purposes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: october 2024-october 2034